CLINICAL TRIAL: NCT00808028
Title: A Randomized, Single-blind, Placebo-controlled, Phase 2 Trial Of The Safety, Immunogenicity, And Tolerability Of Meningococcal Serogroup B (Mnb) Rlp2086 Vaccine At Doses Of 60 Mug, 120 Mug, And 200 Mug In Healthy Adolescents Aged 11 To 18 Years
Brief Title: A Study Evaluating Safety And Immunogenicity Of Meningococcal B Rlp2086 Vaccine In Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6108A1-2001; B1971005 (Other: Alias Study Number); 2008-007789-51 (EudraCT Number)
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Meningitis, Meningococcal
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): dose level 1 rLP2086 vaccine
  Interventions: Biological: meningococcal B rLP2086 vaccine.
- 2 (Experimental): dose level 2 rLP2086 vaccine
  Interventions: Biological: meningococcal B rLP2086 vaccine.
- 3 (Experimental): dose level 3 rLP2086 vaccine
  Interventions: Biological: meningococcal B rLP2086 vaccine.
- 4 (Placebo Comparator): normal saline (placebo)
  Interventions: Other: normal saline (placebo)

INTERVENTIONS:
Biological: meningococcal B rLP2086 vaccine. — vaccine, 0.5 mL, 0 - 2 - 6 to 9 months
  Arms: 1
Biological: meningococcal B rLP2086 vaccine. — vaccine, 0.5 mL, 0 - 2 - 6 to 9 months
  Arms: 2
Biological: meningococcal B rLP2086 vaccine. — vaccine, 0.5 mL, 0 - 2 - 6 to 9 months
  Arms: 3
Other: normal saline (placebo) — vaccine, 0.5 mL, 0 - 2 - 6 to 9 months
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of an investigational meningococcal B rLP2086 vaccine in adolescents aged 11 to 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of >=11 and <=18 years at the time of enrollment.
* Negative urine pregnancy test for all female subjects.
* Parent/legal guardian or subject under supervision of the parent/legal guardian must be able to complete all relevant study procedures during study participation.

Exclusion Criteria:

* History of any invasive meningococcal disease.
* A previous anaphylactic or severe vaccine-associated adverse reaction.
* Any clinically significant chronic disease.
* A known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids. Topical, inhaled or intra-articular corticosteroids are allowed.
* Participation in another investigational study in the 1-month (30-day) period before study visit 1 and during the conduct of the study.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 538 (Actual)
Dates: Start 2009-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Australia (4):
  - Queensland Paediatric Infectious Diseases (QPID) Laboratory, Herston, Queensland
  - Department of Paediatrics, Women's & Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Carlton, Victoria
  - Children's Clinical Research Facility, Vaccine Trials Group (VTG),, Subiaco, Western Australia
- Poland (16):
  - ZOZ w Debicy, Poradnia Chorob Zakaznych, Dębica
  - SP ZOZ Krakowski Szpital Specjalistyczny im. Jana Pawla II w Krakowie, Krakow
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im. Sw. Ludwika w Krakowie,, Krakow
  - Wojewodzki Specjalistyczny Szpital im. dr Wl. Bieganskiego w Lodzi, Lodz
  - Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego, Lodz
  - SPZOZ w Lubartowie, Oddzial Pediatryczny, ul. Cicha 14, Lubartów
  - Eskulap Sp. z o. o., ul. Weteranow 46, Lublin
  - SP ZOZ, Poradnia Dziecieca w Grucie, Mełno
  - NZOZ Pratyka Lekarza Rodzinnego Alina Grocka-Wlazlak, Oborniki Śląskie
  - Specjalistyczny ZOZ nad Matka i Dzieckiem w Poznaniu Oddzial Obserwacyjno-Zakazny A, Poznan
  - NZLA Michalkowice, Jarosz i Partnerzy, Siemianowice Śląskie
  - NZOZ Nasz Lekarz Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia, Torun
  - Oddzial Dzieciecy Szpital im. Swietej Jadwigi Slaskiej, Trzebnica
  - Klinika Pediatrii i Chorob Infekcyjnych, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Wroclaw
  - NZOZ Salmed, Łęczna
- Spain (7):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, La Coruna
  - Hospital U. de Getafe, Getafe, Madrid
  - Hospital U. 12 de Octubre, Madrid, Madrid
  - Complexo Hospitalario Xeral-Cies de Vigo, Vigo, Pontevedra
  - Clinica Virgen del Mar, Almería
  - Hospital General de Cataluna, Barcelona
  - Centro de Salud Nazaret, Valencia

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Beeslaar J, Peyrani P, Absalon J, Maguire J, Eiden J, Balmer P, Maansson R, Perez JL. Sex, Age, and Race Effects on Immunogenicity of MenB-FHbp, A Bivalent Meningococcal B Vaccine: Pooled Evaluation of Clinical Trial Data. Infect Dis Ther. 2020 Sep;9(3):625-639. doi: 10.1007/s40121-020-00322-5. Epub 2020 Jul 17. PMID 32681472
- [Derived] Marshall HS, Richmond PC, Beeslaar J, Jiang Q, Jansen KU, Garces-Sanchez M, Martinon-Torres F, Szenborn L, Wysocki J, Eiden J, Harris SL, Jones TR, Lee SS, Perez JL; 6108A12001 Study Investigators. Meningococcal serogroup B-specific responses after vaccination with bivalent rLP2086: 4 year follow-up of a randomised, single-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2017 Jan;17(1):58-67. doi: 10.1016/S1473-3099(16)30314-0. Epub 2016 Oct 11. PMID 27745812
- [Derived] Richmond PC, Marshall HS, Nissen MD, Jiang Q, Jansen KU, Garces-Sanchez M, Martinon-Torres F, Beeslaar J, Szenborn L, Wysocki J, Eiden J, Harris SL, Jones TR, Perez JL; 2001 Study Investigators. Safety, immunogenicity, and tolerability of meningococcal serogroup B bivalent recombinant lipoprotein 2086 vaccine in healthy adolescents: a randomised, single-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2012 Aug;12(8):597-607. doi: 10.1016/S1473-3099(12)70087-7. Epub 2012 May 7. PMID 22569484
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6108A1-2001&StudyName=A%20Study%20Evaluating%20Safety%20And%20Immunogenicity%20Of%20Meningococcal%20B%20Rlp2086%20Vaccine%20In%20Adolescents

RESULTS

PARTICIPANT FLOW:
Groups:
- Control; rLP2086 120 mcg; rLP2086 200 mcg: Given on a 0, 2-, 6-month schedule in Stage 1 and follow-up to 48 months in Stage 2.
- rLP2086 60 Microgram (mcg): Given on a 0, 2-, 6-month schedule in Stage 1
Period: Stage 1 (6 Months)
Arm/Group | Control | rLP2086 60 Microgram (mcg) | rLP2086 120 mcg | rLP2086 200 mcg
Started | 121 | 22 (Participants in rLP2086 60 mcg group participated only in Stage 1 and were not eligible for Stage 2) | 198 | 198
Completed | 116 | 21 (Participants in rLP2086 60 mcg group participated only in Stage 1 and were not eligible for Stage 2) | 191 | 183
Not Completed | 5 | 1 | 7 | 15
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 5
Not completed — Other | 1 | 0 | 2 | 4
Not completed — Parent/legal guardian request | 0 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Period: Stage 2 (Followed up to 48 Months )
Arm/Group | Control | rLP2086 60 Microgram (mcg) | rLP2086 120 mcg | rLP2086 200 mcg
Started | 80 (Out of 511 completed participants in Stage 1, 89 did not enter Stage 2) | 0 | 170 | 151
Completed | 69 (Out of 511 completed participants in Stage 1, 89 did not enter Stage 2) | 0 | 141 | 128
Not Completed | 11 | 0 | 29 | 23
Not completed — Withdrawal by Subject | 6 | 0 | 9 | 11
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 8 | 7
Not completed — Failed to return | 2 | 0 | 5 | 4
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 1
Not completed — Parent's or guardian request | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The stage 1 intent-to-treat (ITT) population included all randomized participants who received at least 1 vaccination and have at least 1 valid and determinate assay result from blood samples drawn during stage 1.
Groups:
- rLP2086 60 mcg: Given on a 0, 2-, 6-month schedule in Stage 1.
- Total: Total of all reporting groups
Arm/Group | Control | rLP2086 60 mcg | rLP2086 120 mcg | rLP2086 200 mcg | Total
Number analyzed (Participants) | 121 | 22 | 198 | 198 | 539
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.8 (2.05) | 13.3 (1.84) | 14.3 (2.11) | 14.0 (2.01) | 14.0 (2.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 11 | 113 | 103 | 288
  Male | 60 | 11 | 85 | 95 | 251

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 4-fold Rise in Recombinant Lipoprotein 2086 (rLP2086) Specific Serum Bactericidal Assay Using Human Complement (hSBA) Titer: Before Vaccination 1 up to 1 Month After Vaccination 2
Time Frame: Before vaccination 1 up to 1 month after vaccination 2
Population: mITT population included all randomized participants who received at least 1 vaccination and had at least 1 valid and determinate assay result. Here, 'N' signifies those participants who were evaluable for this measure during specified time period.
Measure: Number; unit: Percentage of participants
Groups:
- Control-Stage 1; rLP2086 120 mcg- Stage 1; rLP2086 200 mcg- Stage 1: Given on a 0, 2-, 6-month schedule in Stage 1 and follow-up to 48 months in Stage 2.
- rLP2086 60 mcg- Stage 1: Given on a 0, 2-, 6-month schedule in Stage 1
Arm/Group | Control-Stage 1 | rLP2086 60 mcg- Stage 1 | rLP2086 120 mcg- Stage 1 | rLP2086 200 mcg- Stage 1
Number analyzed (Participants) | 119 | 22 | 195 | 192
Percentage of participants
  Subfamily A Strain A05 (N= 80, 18, 115, 106) | 1.3 | 88.9 | 83.5 | 87.7
  Subfamily B Strain B02 (N= 84, 21, 121, 114) | 0.0 | 71.4 | 59.5 | 59.6
Statistical Analysis 1: Comparison: Control-Stage 1; Strain A05: Response rate was compared with whether greater than (>) 50% of participants had fold rise >=4 using right one-sided exact test based on binomial distribution and the corresponding p-values were calculated. p-value < 0.025 was considered significant; Test type: Superiority or Other; p > 0.9999, Binomial Distribution
Statistical Analysis 2: Comparison: rLP2086 60 mcg- Stage 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0007, Binomial Distribution
Statistical Analysis 3: Comparison: rLP2086 120 mcg- Stage 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial Distribution
Statistical Analysis 4: Comparison: rLP2086 200 mcg- Stage 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial Distribution
Statistical Analysis 5: Comparison: Control-Stage 1; Strain B02: Response rate was compared with whether greater than (>) 50% of participants had fold rise >=4 using right one-sided exact test based on binomial distribution and the corresponding p-values were calculated. p-value < 0.025 was considered significant; Test type: Superiority or Other; p > 0.9999, Binomial Distribution
Statistical Analysis 6: Comparison: rLP2086 60 mcg- Stage 1; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.0392, Binomial Distribution
Statistical Analysis 7: Comparison: rLP2086 120 mcg- Stage 1; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.0225, Binomial Distribution
Statistical Analysis 8: Comparison: rLP2086 200 mcg- Stage 1; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.0244, Binomial Distribution

2. Primary Outcome: Percentage of Participants With at Least 4-fold Rise in Recombinant Lipoprotein 2086 (rLP2086) Specific Serum Bactericidal Assay Using Human Complement (hSBA) Titer: Before Vaccination 1 up to 1 Month After Vaccination 3
Time Frame: Before vaccination 1 up to 1 month after vaccination 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Control-Stage 1 | rLP2086 60 mcg- Stage 1 | rLP2086 120 mcg- Stage 1 | rLP2086 200 mcg- Stage 1
Number analyzed (Participants) | 119 | 22 | 195 | 192
Percentage of participants
  Subfamily A Strain A05 (N= 73, 19, 111,100) | 5.5 | 89.5 | 92.8 | 94.0
  Subfamily B Strain B02 (N= 79, 21, 112,105) | 1.3 | 81.0 | 86.6 | 84.8
Statistical Analysis 1: Comparison: Control-Stage 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.9999, Binomial Distribution
Statistical Analysis 2: Comparison: rLP2086 60 mcg- Stage 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0004, Binomial Distribution
Statistical Analysis 3: Comparison: rLP2086 120 mcg- Stage 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial Distribution
Statistical Analysis 4: Comparison: rLP2086 200 mcg- Stage 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial Distribution
Statistical Analysis 5: Comparison: Control-Stage 1; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p > 0.9999, Binomial Distribution
Statistical Analysis 6: Comparison: rLP2086 60 mcg- Stage 1; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.0036, Binomial Distribution
Statistical Analysis 7: Comparison: rLP2086 120 mcg- Stage 1; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p < 0.0001, Binomial Distribution
Statistical Analysis 8: Comparison: rLP2086 200 mcg- Stage 1; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p < 0.0001, Binomial Distribution

3. Primary Outcome: Percentage of Participants With Atleast One Adverse Event (AE): Stage 1
Time Frame: Vaccination 1 upto 1 Month after vaccination 3
Population: Safety population included participants who received at least 1 dose of study vaccine.
Measure: Number; unit: Percentage of participants
Arm/Group | Control-Stage 1 | rLP2086 60 mcg- Stage 1 | rLP2086 120 mcg- Stage 1 | rLP2086 200 mcg- Stage 1
Number analyzed (Participants) | 121 | 22 | 198 | 195
Percentage of participants
  Stage 1: Vaccination phase | 44.6 | 81.8 | 38.9 | 47.2
  Stage 1: 6-month follow up phase | 4.1 | 18.2 | 1.5 | 2.6

4. Primary Outcome: Percentage of Participants With Atleast One Adverse Event (AE): Stage 2
Time Frame: 6 month after vaccination 3 up to 48 months
Population: Safety population included participants who received at least 1 dose of study vaccine.
Measure: Number; unit: Percentage of participants
Groups:
- Control- Stage 2; rLP2086 120 mcg- Stage 2; rLP2086 200 mcg- Stage 2: Given on a 0, 2-, 6-month schedule in Stage 1, were then followed up to 48 months in Stage 2.
Arm/Group | Control- Stage 2 | rLP2086 120 mcg- Stage 2 | rLP2086 200 mcg- Stage 2
Number analyzed (Participants) | 80 | 170 | 151
Percentage of participants | 2.5 | 4.1 | 2.0

5. Secondary Outcome: Percentage of Participants Achieving Serum Bactericidal Assay Using Human Complement (hSBA) Titer Level Greater Than or Equal To (>=) Prespecified Titer Level
Time Frame: 1 month before vaccination 1, 1 month after vaccination 2, 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Control-Stage 1 | rLP2086 60 mcg- Stage 1 | rLP2086 120 mcg- Stage 1 | rLP2086 200 mcg- Stage 1
Number analyzed (Participants) | 119 | 22 | 195 | 192
Percentage of participants
  A04 Predose 1;1:32 (N= 64, 15, 90, 92) | 10.9 | 0.0 | 10.0 | 12.0
  A04 Predose 1;1:64 (N= 64, 15, 90, 92) | 3.1 | 0.0 | 7.8 | 5.4
  A04 Predose 1;1:128 (N= 64, 15, 90, 92) | 0.0 | 0.0 | 1.1 | 0.0
  A04 1-month postdose 2;1:32 (N= 69, 21, 115, 115) | 4.3 | 95.2 | 98.3 | 91.3
  A04 1-month postdose 2;1:64 (N= 69, 21, 115, 115) | 1.4 | 85.7 | 82.6 | 72.2
  A04 1-month postdose 2;1:128 (N= 69, 21, 115, 115) | 1.4 | 52.4 | 44.3 | 42.6
  A05 Predose 1;1:16 (N= 81, 21, 122, 114) | 12.3 | 4.8 | 9.0 | 6.1
  A05 Predose 1;1:32 (N= 81, 21, 122, 114) | 7.4 | 4.8 | 5.7 | 4.4
  A05 Predose 1;1:64 (N= 81, 21, 122, 114) | 4.9 | 0.0 | 2.5 | 1.8
  A05 Predose 1;1:128 (N= 81, 21, 122, 114) | 1.2 | 0.0 | 0.8 | 0.0
  A05 1-month postdose 2;1:16 (N= 83, 18, 118, 110) | 7.2 | 88.9 | 89.0 | 90.9
  A05 1-month postdose 2;1:32 (N= 83, 18, 118, 110) | 3.6 | 88.9 | 85.6 | 81.8
  A05 1-month postdose 2;1:64 (N= 83, 18, 118, 110) | 1.2 | 83.3 | 59.3 | 64.5
  A05 1-month postdose 2;1:128 (N= 83, 18, 118, 110) | 0.0 | 33.3 | 28.0 | 40.0
  A05 1-month postdose 3;1:16 (N= 76, 20, 114, 104) | 11.8 | 90.0 | 96.5 | 96.2
  A05 1-month postdose 3;1:32 (N= 76, 20, 114, 104) | 7.9 | 90.0 | 94.7 | 95.2
  A05 1-month postdose 3;1:64 (N= 76, 20, 114, 104) | 3.9 | 85.0 | 89.5 | 87.5
  A05 1-month postdose 3;1:128 (N= 76, 20, 114, 104) | 1.3 | 40.0 | 68.4 | 60.6
  A56 Predose 1;1:16 (N= 80, 21, 119, 115) | 10.0 | 4.8 | 7.6 | 6.1
  A56 Predose 1;1:32 (N= 80, 21, 119, 115) | 7.5 | 4.8 | 5.0 | 4.3
  A56 Predose 1;1:64 (N= 80, 21, 119, 115) | 2.5 | 0.0 | 0.8 | 3.5
  A56 Predose 1;1:128 (N= 80, 21, 119, 115) | 1.3 | 0.0 | 0.0 | 0.0
  A56 1-month postdose 2;1:16 (N= 81, 20, 117, 107) | 12.3 | 85.0 | 94.9 | 96.3
  A56 1-month postdose 2;1:32 (N= 81, 20, 117, 107) | 11.1 | 85.0 | 90.6 | 88.8
  A56 1-month postdose 2;1:64 (N= 81, 20, 117, 107) | 9.9 | 80.0 | 80.3 | 71.0
  A56 1-month postdose 2;1:128 (N= 81, 20, 117, 107) | 2.5 | 45.0 | 39.3 | 45.8
  A56 1-month postdose 3 ;1:16 (N= 78, 21, 114, 112) | 11.5 | 95.2 | 97.4 | 95.5
  A56 1-month postdose 3 ;1:32 (N= 78, 21, 114, 112) | 9.0 | 85.7 | 93.9 | 93.8
  A56 1-month postdose 3 ;1:64 (n= 78, 21, 114, 112) | 3.8 | 71.4 | 91.2 | 84.8
  A56 1-month postdose 3;1:128 (N= 78, 21, 114, 112) | 2.6 | 61.9 | 74.6 | 67.0
  B02 postdose 1;1:16 (N= 84, 22, 124, 118) | 3.6 | 0.0 | 1.6 | 2.5
  B02 postdose 1;1:32 (N= 84, 22, 124, 118) | 1.2 | 0.0 | 0.8 | 1.7
  B02 postdose 1;1:64 (N= 84, 22, 124, 118) | 0.0 | 0.0 | 0.8 | 0.0
  B02 postdose 1;1:128 (N= 84, 22, 124, 118) | 0.0 | 0.0 | 0.8 | 0.0
  B02 1-month postdose 2 ;1:16 (N= 84, 21, 122, 114) | 1.2 | 76.2 | 68.9 | 65.8
  B02 1-month postdose 2 ;1:32 (N= 84, 21, 122, 114) | 0.0 | 57.1 | 45.9 | 48.2
  B02 1-month postdose 2 ;1:64 (N= 84, 21, 122, 114) | 0.0 | 42.9 | 25.4 | 21.9
  B02 1-month postdose 2;1:128 (N= 84, 21, 122, 114) | 0.0 | 14.3 | 7.4 | 8.8
  B02 1-month postdose 3 ;1:16 (N= 79, 21, 113, 105) | 3.8 | 85.7 | 90.3 | 85.7
  B02 1-month postdose 3 ;1:32 (N= 79, 21, 113, 105) | 1.3 | 81.0 | 78.8 | 79.0
  B02 1-month postdose 3 ;1:64 (N= 79, 21, 113, 105) | 0.0 | 57.1 | 52.2 | 60.0
  B02 1-month postdose 3;1:128 (N= 79, 21, 113, 105) | 0.0 | 42.9 | 19.5 | 19.0
  B03 Predose 1;1:16 (N= 83, 22, 118, 117) | 2.4 | 0.0 | 2.5 | 2.6
  B03 Predose 1;1:32 (N= 83, 22, 118, 117) | 2.4 | 0.0 | 2.5 | 2.6
  B03 Predose 1;1:64 (N= 83, 22, 118, 117) | 1.2 | 0.0 | 0.0 | 0.9
  B03 Predose 1;1:128 (N= 83, 22, 118, 117) | 0.0 | 0.0 | 0.0 | 0.0
  B03 1-month postdose 2;1:16 (N= 84, 19, 102, 96) | 2.4 | 21.1 | 32.4 | 30.2
  B03 1-month postdose 2;1:32 (N= 84, 19, 102, 96) | 2.4 | 21.1 | 30.4 | 28.1
  B03 1-month postdose 2;1:64 (N= 84, 19, 102, 96) | 1.2 | 5.3 | 22.5 | 19.8
  B03 1-month postdose 2;1:128 (N= 84, 19, 102, 96) | 0.0 | 0.0 | 10.8 | 2.3
  B03 1-month postdose 3;1:16 (N= 68, 15, 86, 81) | 5.9 | 53.3 | 75.6 | 67.9
  B03 1-month postdose 3;1:32 (N= 68, 15, 86, 81) | 4.4 | 53.3 | 75.6 | 66.7
  B03 1-month postdose 3;1:64 (N= 68, 15, 86, 81) | 1.5 | 46.7 | 60.5 | 58.0
  B03 1-month postdose 3;1:128 (N= 68, 15, 86, 81) | 0.0 | 26.7 | 27.9 | 24.7
  B44 Predose 1 ;1:8 (N= 81, 22, 120, 116) | 2.5 | 0.0 | 3.3 | 2.6
  B44 Predose 1 ;1:16 (N= 81, 22, 120, 116) | 1.2 | 0.0 | 1.7 | 2.6
  B44 Predose 1 ;1:32 (N= 81, 22, 120, 116) | 0.0 | 0.0 | 0.0 | 1.7
  B44 Predose 1 ;1:64 (N= 81, 22, 120, 116) | 0.0 | 0.0 | 0.0 | 0.9
  B44 Predose 1 ;1:128 (N= 81, 22, 120, 116) | 0.0 | 0.0 | 0.0 | 0.9
  B44 1-month postdose 2;1:8 (n= 81, 21, 115, 106) | 1.2 | 61.9 | 68.7 | 70.8
  B44 1-month postdose 2;1:16 (N= 81, 21, 115, 106) | 0.0 | 61.9 | 60.9 | 64.2
  B44 1-month postdose 2;1:32 (N= 81, 21, 115, 106) | 0.0 | 47.6 | 43.5 | 42.5
  B44 1-month postdose 2;1:64 (N= 81, 21, 115, 106) | 0.0 | 23.8 | 22.6 | 25.5
  B44 1-month postdose 2;1:128 (N= 81, 21, 115, 106) | 0.0 | 0.0 | 6.1 | 11.3
  B44 1-month postdose 3;1:8 (N= 83, 21, 115, 111) | 4.8 | 76.2 | 88.7 | 86.5
  B44 1-month postdose 3; 1:16 (N= 83, 21, 115, 111) | 1.2 | 76.2 | 86.1 | 85.6
  B44 1-month postdose 3;1:32 (N= 83, 21, 115, 111) | 0.0 | 76.2 | 80.9 | 80.2
  B44 1-month postdose 3;1:64 (N= 83, 21, 115, 111) | 0.0 | 47.6 | 53.9 | 61.3
  B44 1-month postdose 3;1:128 (N= 83, 21, 115, 111) | 0.0 | 9.5 | 22.6 | 19.8

6. Other Pre Specified Outcome: Immunogloblulin G (IgG) Measured by Geometric Mean Titer (GMT) for Sub Family A and Sub Family B
Time Frame: Before Vaccination 1, 1 month after vaccination 2, 1 month after vaccination 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Control-Stage 1 | rLP2086 60 mcg- Stage 1 | rLP2086 120 mcg- Stage 1 | rLP2086 200 mcg- Stage 1
Number analyzed (Participants) | 119 | 22 | 195 | 192
Titer
  Subfamily(Sf) A Predose 1(N=106,22,156,173) | 3.6 [2.6 to 5.1] | 4.3 [1.6 to 11.7] | 7.2 [5.3 to 9.8] | 4.9 [3.8 to 6.4]
  Sf A 1-month postdose 2(N=104, 22,168,166) | 4.9 [3.5 to 6.9] | 984.6 [663.8 to 1460.4] | 1115.5 [962.8 to 1292.5] | 1285.8 [1082.3 to 1527.7]
  Sf A 1-month postdose 3(N=98,20, 158,148) | 5.8 [3.9 to 8.5] | 3120.3 [1959.5 to 4968.8] | 2289.5 [1967.0 to 2664.9] | 2342.6 [2003.9 to 2738.5]
  Sf B Predose 1(N= 106,22,155,172) | 3.5 [2.6 to 4.6] | 4.2 [1.4 to 12.7] | 5.4 [4.1 to 7.2] | 3.9 [3.0 to 5.0]
  Sf B 1-month postdose 2(N=104, 22,168,166) | 3.7 [2.7 to 5.0] | 405.8 [298.7 to 551.4] | 816.5 [701.0 to 951.1] | 852.0 [729.1 to 995.6]
  Sf B 1-month postdose 3(N=98,20,158,148) | 4.1 [2.9 to 5.7] | 3264.2 [2502.3 to 4258.1] | 2246.8 [1988.1 to 2539.2] | 2553.3 [2256.0 to 2889.7]

ADVERSE EVENTS:
Time Frame: AE reported from Vaccination 1 upto 48 months after vaccincation 3 and SAE reported from Vaccination 1 upto 48 months after vaccincation 3
Groups:
- Control- Stage 1; rLP2086 60 mcg- Stage 1; rLP2086 120 mcg- Stage 1; rLP2086 200 mcg- Stage 1: Given on a 0, 2-, 6-month schedule in Stage 1
- Control-Stage 1 Follow-up; rLP2086 60 mcg- Stage 1 Follow up; rLP2086 120 mcg- Stage 1 Follow up; rLP2086 200 mcg- Stage 1 Follow up: Given on a 0, 2-, 6-month schedule in Stage 1, were then followed up to 6 months in Stage 1
- Control-Stage 2; rLP2086 120 mcg- Stage 2; rLP2086 200 mcg- Stage 2: Given on a 0, 2-, 6-month schedule in Stage 1, were then followed up to 6 months in Stage 1 and further up to 48 months in Stage 2
Arm/Group | Control- Stage 1 | rLP2086 60 mcg- Stage 1 | rLP2086 120 mcg- Stage 1 | rLP2086 200 mcg- Stage 1 | Control-Stage 1 Follow-up | rLP2086 60 mcg- Stage 1 Follow up | rLP2086 120 mcg- Stage 1 Follow up | rLP2086 200 mcg- Stage 1 Follow up | Control-Stage 2 | rLP2086 120 mcg- Stage 2 | rLP2086 200 mcg- Stage 2
Serious Adverse Events (participants affected / at risk) | 3/121 | 1/22 | 3/198 | 8/195 | 0/121 | 1/22 | 1/198 | 2/195 | 1/80 | 6/170 | 3/151
Other Adverse Events (participants affected / at risk) | 54/121 | 18/22 | 75/198 | 91/195 | 5/121 | 3/22 | 2/198 | 4/195 | 1/80 | 1/170 | 0/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control- Stage 1 (N=121) | rLP2086 60 mcg- Stage 1 (N=22) | rLP2086 120 mcg- Stage 1 (N=198) | rLP2086 200 mcg- Stage 1 (N=195) | Control-Stage 1 Follow-up (N=121) | rLP2086 60 mcg- Stage 1 Follow up (N=22) | rLP2086 120 mcg- Stage 1 Follow up (N=198) | rLP2086 200 mcg- Stage 1 Follow up (N=195) | Control-Stage 2 (N=80) | rLP2086 120 mcg- Stage 2 (N=170) | rLP2086 200 mcg- Stage 2 (N=151)
Eczema impetiginous (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CNS germinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mononucleosis syndrome (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control- Stage 1 (N=121) | rLP2086 60 mcg- Stage 1 (N=22) | rLP2086 120 mcg- Stage 1 (N=198) | rLP2086 200 mcg- Stage 1 (N=195) | Control-Stage 1 Follow-up (N=121) | rLP2086 60 mcg- Stage 1 Follow up (N=22) | rLP2086 120 mcg- Stage 1 Follow up (N=198) | rLP2086 200 mcg- Stage 1 Follow up (N=195) | Control-Stage 2 (N=80) | rLP2086 120 mcg- Stage 2 (N=170) | rLP2086 200 mcg- Stage 2 (N=151)
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 20 | 13 | 28 | 21 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid cyst (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 4 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site dermatitis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pallor (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site paraesthesia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site pallor (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to chemicals (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 5 | 0 | 4 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 8 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 4 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mumps (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hangnail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation mucosal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.